CLINICAL TRIAL: NCT00874367
Title: Early-Onset Sepsis: an NICHD/CDC Surveillance Study
Brief Title: Early-Onset Sepsis Surveillance Study
Acronym: EOS
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0035; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD036790 (NIH); U10HD040492 (NIH); U10HD040498 (NIH); U10HD040521 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024139 (NIH); UL1RR025744 (NIH); UL1RR025764 (NIH); UL1RR025777 (NIH); M01RR000030 (NIH); M01RR000032 (NIH); M01RR000039 (NIH); M01RR000044 (NIH); M01RR000054 (NIH); M01RR000059 (NIH); M01RR000064 (NIH); M01RR000070 (NIH); M01RR000080 (NIH); M01RR000633 (NIH); M01RR000750 (NIH); M01RR000997 (NIH); M01RR008084 (NIH); M01RR006022 (NIH); M01RR007122 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Sepsis; Gram-Negative Bacterial Infections; Gram-Positive Bacterial Infections
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity; Early Onset Sepsis
MeSH Terms: conditions — Premature Birth; Sepsis; Gram-Negative Bacterial Infections; Gram-Positive Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of the isolated pathogens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this observational study, the NICHD Neonatal Research Network (NRN) is conducting surveillance of all infants born at NRN centers to identify all newborns who are diagnosed with early-onset sepsis (EOS) and/or meningitis. The study will: establish current hospital-based rates of EOS among term and preterm infants in the era of intrapartum antibiotic prophylaxis; monitor the organisms associated with EOS and meningitis; compare asymptomatic and symptomatic infants by gestational age and pathogen; and monitor sepsis-associated mortality rates by pathogen group.

DETAILED DESCRIPTION:
For more than a decade, the NICHD Neonatal Research Network (NRN) has conducted surveillance of early-onset sepsis (EOS) infections in very low birth weight (VLBW) infants, as part of its very low birth weight registry. Although overall rates of EOS have remained stable over time, the relative importance of different pathogens has changed.

In 2002 the American Academy of Pediatrics, the American College of Obstetricians and Gynecologists, and the Centers for Disease Control & Prevention revised their recommendations for reducing mother-to-child transmission of group B streptococcal (GBS) infections. The new guidelines recommend universal screening of pregnant women at 35 or more weeks' gestation and intrapartum antibiotics for all GBS-colonized mothers (an estimated 30% of mother-to-be in the United States). With the current widespread use of maternal antibiotics, concerns have been raised about the possible emergence of non-GBS pathogens as causes of early-onset sepsis. Several studies have reported a change in EOS pathogens, with the emergence of gram-negative and antibiotic-resistant infections, primarily among VLBW infants.

This observational study expands the NRN's prior work on infection in VLBW infants, conducting surveillance of all infants born at network centers who are diagnosed with early-onset sepsis and/or meningitis. The study will: establish current hospital-based rates of EOS among term and preterm infants in the era of intrapartum antibiotic prophylaxis; monitor the organisms associated with EOS and meningitis; compare asymptomatic and symptomatic infants by gestational age and pathogen; and monitor sepsis-associated mortality rates by pathogen group. Cases will be identified by the medical care team or through research team review of patient, microbiology, or infection control/hospital epidemiology records.

Secondary analyses include:

Serotypic, phylogenetic, virulence and drug-resistance characteristics of contemporary GBS and E. Coli isolate collections will be studied.

Assessing the proportion of neonates born to mothers with chorioamnionitis who are asymptomatic at birth, but later develop signs and/or symptoms of early-onset neonatal GBS and non-GBS disease.

ELIGIBILITY:
Inclusion Criteria:

* Infants >400g birth weight

Exclusion Criteria:

* Stillbirth or death in the delivery room

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All live born infants >400g birth weight delivered at NICHD Neonatal Research Network participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Early onset sepsis infections | Until hospital discharge

SECONDARY OUTCOMES:
Group B streptococcal (GBS) infections | Until hospital discharge
Symptomatic early onset sepsis infections | Until hospital discharge
Death with early gram-negative or early gram-positive infections | Until hospital discharge
Prolonged exposure to maternal intrapartum antibiotics (>24 hours) | Prenatal
Placental examinations to confirm clinical diagnosis of chorioamnionitis | Prenatal

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Frantz III, MD, Principal Investigator — Tufts Medical Center; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Bell, MD, Principal Investigator — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Roger G. Faix, MD, Principal Investigator — University of Utah; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Dale L. Phelps, MD, Principal Investigator — University of Rochester; T. Michael O'Shea, MD, Principal Investigator — Wake Forest University
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Stoll BJ, Hansen NI, Sanchez PJ, Faix RG, Poindexter BB, Van Meurs KP, Bizzarro MJ, Goldberg RN, Frantz ID 3rd, Hale EC, Shankaran S, Kennedy K, Carlo WA, Watterberg KL, Bell EF, Walsh MC, Schibler K, Laptook AR, Shane AL, Schrag SJ, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Early onset neonatal sepsis: the burden of group B Streptococcal and E. coli disease continues. Pediatrics. 2011 May;127(5):817-26. doi: 10.1542/peds.2010-2217. Epub 2011 Apr 25. PMID 21518717
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/